CLINICAL TRIAL: NCT01943669
Title: An Open, Longitudinal, Prospective, Non-randomized, Self-Controlled Feasibility Study to Investigate the Effect of the ReWalk™ Device on Mobility Outcomes in Patients With Chronic Spinal Cord Injury.
Brief Title: Exoskeletons for Spinal Cord Injury: A Feasibility Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Buckinghamshire Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 13/EE/0048 (UK NRES)
Record Dates: First submitted 2013-07-22; First posted 2013-09-17 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2013-09

CONDITIONS: Spinal Cord Injury
Keywords: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Exoskeleton Device

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ReWalk™ device (Experimental): Self-controlled group; single cohort.
  Interventions: Device: ReWalk™ device

INTERVENTIONS:
Device: ReWalk™ device — Twenty one-hour ReWalk™ training sessions are scheduled for each participant over a 10-week period.
  Other Names: Exoskeleton; Bionic suit

SUMMARY:
In this study, 10 volunteer participants with chronic spinal cord injury will undergo a 10-week training schedule for ambulation with the ReWalk™ device. The ReWalk™ consists of a lightweight brace-support suit containing motors at the hip and knee joints, rechargeable batteries and a computerized control system carried in a backpack. ReWalk™ users control their ambulation through subtle changes in centre of gravity and upper-body movements. Before, during and after training sessions the volunteers will perform standardised assessments and complete questionnaires to assess the functional and psychological effects of the exoskeleton. Functional outcomes primarily focus on ambulation outcomes and psychological outcomes primarily focus on predisposition and perceptions of disability. The outcomes of this pilot study will assist the investigators in the preparations of randomised controlled trail for assessing the efficacy of the ReWalk™ device in a neurorehabilitation setting.

DETAILED DESCRIPTION:
In this study, 10 volunteer participants with chronic spinal cord injury will undergo a 10-week training schedule for ambulation with the ReWalk™ device. The ReWalk™ consists of a lightweight brace-support suit containing motors at the hip and knee joints, rechargeable batteries and a computerized control system carried in a backpack. ReWalk™ users control their ambulation through subtle changes in centre of gravity and upper-body movements. Before, during and after training sessions the volunteers will perform standardised assessments and complete questionnaires to assess the functional and psychological effects of the exoskeleton. Twenty one-hour training sessions are scheduled for each participant over a 10-week period. Functional outcomes primarily focus on ambulation outcomes and psychological outcomes primarily focus on predisposition and perceptions of disability. The outcomes of this pilot study will assist the investigators in the preparations of randomised controlled trail for assessing the efficacy of the ReWalk™ device in a neurorehabilitation setting.

ELIGIBILITY:
Inclusion Criteria:

* American Spinal Injury Association (ASIA) Impairment Scale (AIS) grade A, B & C (Lower Extremity Motor Score <20)
* Motor level of injury from Cervical level 7 to Lumbar level 1, according to ASIA guidelines
* Male and non-pregnant, non-lactating female
* Age 18-55 years old
* At least 12 months after injury
* Able to stand or maintain upright position with or without using a standing device (e.g., 'Easy stand')
* Able to sit with hips and knees ≥90° flexion
* Height of 160 to 190 cm
* Weight of <100 kg

Exclusion Criteria:

* History of severe neurological injuries other than spinal cord injury (eg. Multiple Sclerosis, Cerebral Palsy, Amyotrophic Lateral Sclerosis, Traumatic Brain Injury, Stroke)
* Concurrent medical diseases (eg. infections, circulatory, heart or lung, pressure sores) interfering with the study
* Unstable spine or unhealed limbs or pelvic fractures
* Limited range of motion (<90°) hip and knee joints, including severe contractures
* Severe spasticity (Ashworth grade 4; ie. Affected part(s) rigid in flexion or extension) or uncontrolled clonus
* Diagnosis of severe osteoporosis/penia as proven with pQCT or DXA.
* Psychiatric or cognitive conditions that may interfere with the trial
* Previous use of any exoskeletal robotic device
* Patients incapable of providing informed consent

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2013-06; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
10-meter walking test (10MWT) | 10 weeks
  Change in score between 0 and 10 weeks.

SECONDARY OUTCOMES:
6-minutes walk test (6MWT) | 10 weeks
  Change in score between 0 and 10 weeks.
Timed Up and Go (TUG) test | 10 weeks
  Change in score between 0 and 10 weeks.
Assistive Technology Device Predisposition Assessment© (ATDPA) Questionnaire | 10 weeks
  Change in score between 0 and 10 weeks.
Appraisals of Disability: Primary and Secondary Scale (ADAPSS) Questionnaire | 10 weeks
  Change in score between 0 and 10 weeks.

OTHER OUTCOMES:
Stair management | 10 weeks
  Exact timing pending learning curve, change in score in weeks up to 10 weeks.
Obstacle course | 10 weeks
  Exact timing pending learning curve, change in score in weeks up to 10 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Joost J. van Middendorp, MD, PhD, Principal Investigator — Stoke Mandeville Spinal Foundation
Locations (1):
- National Spinal Injuries Centre, Stoke Mandeville Hospital, Aylesbury, Buckinghamshire, United Kingdom

REFERENCES:
- See also: Website directing to project description and updates — http://www.smsf.org.uk/research%20introduction.htm